CLINICAL TRIAL: NCT00258206
Title: Phase II Study of High Dose Cyclophosphamide and Rituximab in Multiple Myeloma
Brief Title: Rituximab and Cyclophosphamide in Treating Patients With High Risk, Refractory, or Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0478 CDR0000441169; P30CA006973 (NIH); JHOC-J0478 (Other: Johns Hopkins SKCCC)
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Results first posted 2015-06-11 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Rituximab; Cyclophosphamide

ARMS (1):
- rituximab + cyclophosphamide (Experimental): Rituximab 375 mg/m^2 on Days -10 and -7; Cyclophosphamide 50 mg/kg on days -3, -2, -1, and 0; Rituximab 375 mg/m^2 weekly x4 after platelet counts recover; For patients achieving at least stable disease, rituximab maintenance 375 mg/m^2 once each during months 3, 6, 9, and 12
  Interventions: Biological: rituximab; Drug: cyclophosphamide

INTERVENTIONS:
Biological: rituximab
  Other Names: Rituxan
Drug: cyclophosphamide
  Other Names: Cytoxan

SUMMARY:
RATIONALE: Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving rituximab together with cyclophosphamide may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving rituximab together with cyclophosphamide works in treating patients with high risk, refractory, or relapsed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of rituximab and high-dose cyclophosphamide on the growth of myeloma stem cells in patients with high-risk, refractory, or relapsed multiple myeloma.

OUTLINE: Patients receive rituximab IV on days -10 and -7; once weekly for 4 weeks (after completion of high-dose cyclophosphamide); and then once in months 3, 6, 9, and 12. Patients also receive high-dose cyclophosphamide on days -3 to 0.

PROJECTED ACCRUAL: Not specified.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma, meeting 1 of the following criteria:

  * High-risk disease in first remission, as defined by the following:

    * Beta-2 microglobulin > 5.0 mg/dL
    * Chromosome 13 deletion
  * Primary refractory disease
  * Relapsed disease after achieving a response to prior chemotherapy
* The following diagnoses are not allowed:

  * POEMS syndrome
  * Plasma cell leukemia
  * Amyloidosis
  * Nonsecretory myeloma
* No evidence of spinal cord compression

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* Has good organ function
* Is in good physical condition
* No active infection requiring antibiotics
* No other malignancy within the past 2 years except basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No persistently detectable donor cells after prior allogeneic stem cell transplantation
* No prior rituximab

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 28 days since prior therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2004-12; Primary Completion 2007-09-07 (Actual); Study Completion 2007-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carol A. Huff, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab + Cyclophosphamide
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab + Cyclophosphamide
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Percentage of study participants who did not report that their multiple myeloma relapsed or progressed (got worse)
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab + Cyclophosphamide
Number analyzed (Participants) | 21
percentage of participants | 29

2. Primary Outcome: Safety of Maintenance Rituximab Following High Dose Cyclophosphamide
Time Frame: 2, 3, 6, 9, and 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Safety and Toxicity
Time Frame: 2, 3, 6, 9, and 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Complete Response (CR) Rate and Partial Response (PR) Rate
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: Effect of Rituximab by Clonogenic Growth of Multiple Myeloma (MM) Progenitors and the Mechanisms by Which MM Stem Cells Are Inhibited
Time Frame: 2, 3, 6, 9, and 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Rituximab + Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes